CLINICAL TRIAL: NCT04752995
Title: Proximal Tibial Osteotomy Osteoclasis In Infantile Genu-Varum: Improving the Technique and Managing Potential Complications.
Brief Title: Proximal Tibial Osteotomy Osteoclasis In Infantile Genu-Varum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ahmed m. samy, assisstant professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tanta u
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Deformity Knee; Deformity of Limb
Keywords: Genu varum, mini-invasive, osteotomy, osteoclasis
MeSH Terms: conditions — Genu Varum | interventions — Osteotomy

STUDY DESIGN:
Intervention Model Description: prospective randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high tibial osteotomy (Other): Under general anesthesia, a one-cm vertical skin incision was done at the medial subcutaneous border of the tibia, one fingerbreadth below the tibial tuberosity. This was confirmed by intra-operative C-arm images. Longitudinal periosteal incision was done with minimal dissection. Incomplete medial transverse osteotomy including both anterior and posterior cortex was performed using drill bit or small thin osteotome.Osteotomy was completed manually by osteoclasis of the lateral cortex to provide postoperative stability by the preserved lateral periosteum. No fibular osteotomy was needed in the present study.
  Interventions: Procedure: osteotomy

INTERVENTIONS:
Procedure: osteotomy — osteotomy osteoclasis of upper tibia

SUMMARY:
Genu-varum is a common problem encountered in pediatric orthopedic. Correction of pathological deformity is mandatory to ensure normal load transfer through the knee. In this study, the investigators describe a new technique of osteotomy osteoclasis in order to evaluate if it is an effective and reliable method in management of infantile genu varum

DETAILED DESCRIPTION:
Seventy children with 122 legs suffering significant infantile genu-varum were treated by percutaneous osteotomy-osteoclasis technique. The mean age was 46 months. Genu varum was bilateral in 52 children and unilateral in 18 with a mean preoperative proximal medial tibial angle 66.67 ± 2.670. Under general anesthesia, transverse osteotomy osteoclasis was performed below the tibial tuberosity. Follow-up radiograph was done within the first post-operative week and then every two weeks to assess alignment and consolidation.

ELIGIBILITY:
Inclusion criteria:

* Infantile genu-varum
* PMTA≤70 not spontaneously corrected

Exclusion criteria:

* Active rickets or other metabolic disease
* Patients in whom the femur or the joint is the main site of the deformity

Ages: 36 Months to 52 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
proximal medial tibial angle | one year
  This angle was used for assessment of degree of deformity correction and to follow the presence of under- or over-correction
the posterior proximal tibial angle | one year
  confirm the absence or presence of any sagittal pro or recurvatum deformities(normal=81±2 degrees)
Self-Administered Patient Satisfaction Scale | one year
  the investigators asked the parents to rate their satisfaction on a scale from zero to 100 (100 to 75 very satisfied, <75 to 50 somewhat satisfied, <50 to 25 somewhat dissatisfied and <25 dissatisfied).Those who were not satisfied are requested to explain the cause of dissatisfaction.

IPD SHARING:
Plan to Share IPD: No
the investigators will publish the final results

REFERENCES:
- [Background] Rab GT. Oblique tibial osteotomy revisited. J Child Orthop. 2010 Apr;4(2):169-72. doi: 10.1007/s11832-009-0228-z. Epub 2009 Dec 20. PMID 20234769